CLINICAL TRIAL: NCT06246318
Title: Effects of Virtual Reality in Children With Developmental Coordination Disorder: Randomized Controlled Trial
Brief Title: Effects of VR in Children With DCD: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ZEYNEP KOLİT, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR24
Record Dates: First submitted 2024-01-17; First posted 2024-02-07 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Virtual Reality; Developmental Coordination Disorder; Visual Perceptual Weakness; Motor Skills Disorders; Sensory Disorder; Executive Dysfunction; Participation, Patient
Keywords: virtual reality; Visual Perceptual; motor skills; Developmental Coordination Disorder; sensory perception; cognition; participation
MeSH Terms: conditions — Motor Skills Disorders; Sensation Disorders; Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality plus conventional occupational therapy (Experimental): Virtual reality will be given to the study group in addition to the conventional occupational therapy program.
  Nintendo Wii Fit Plus will be used as the virtual reality method in the research.
  Interventions: Other: virtual reality; Other: conventional occupational therapy
- conventional occupational therapy (Other): This is a control group. Sensory integration and gross motor training approaches are used in the conventional occupational therapy program.
  Interventions: Other: conventional occupational therapy

INTERVENTIONS:
Other: virtual reality — The virtual reality protocol here is based on perceptual-motor activities, supported by Nintendo Wii resources. The user will be able to control a game character in a virtual environment using a remote control with a motion sensor. Wii Fit Plus requires the use of the Wii Balance Board that the player stands on during gameplay. The Wii Balance Board is not a wobbly balance board, but is able to detect and track the user's center of balance, a feature used extensively in the game. Wii Fit Plus includes more than 40 activities including yoga, strength training, aerobics and balance games. During the virtual reality application, different games will be preferred in each session depending on the duration of the games. Virtual reality application will be carried out in a corner prepared for virtual reality application in the room where the conventional occupational therapy session is held. Families have the right to observe and attend all sessions whenever they wish.
  Arms: virtual reality plus conventional occupational therapy
Other: conventional occupational therapy — Sensory integration and gross motor training approaches will be used in the conventional occupational therapy program. A manualized protocol based on Ayres sensory integration principles will be followed (Schaaf et al., 2012). The intervention will be carried out by a licensed occupational therapist trained in sensory integration.
  This approach suggests that if a child engages in individually adapted sensorimotor activities, the nervous system is better able to modulate, organize, and integrate sensory information and is also more likely to use sensory information in adaptive ways (Ayres, 1972). Components of the intervention include a sensory-rich, playful, child-centered approach, providing a decision challenge, and facilitating increasingly complex adaptive behaviors by engaging the child in individually tailored, developmentally appropriate play interactions

SUMMARY:
The aim of the study is to examine the effect of VR application on motor, cognitive and sensory-perceptual skills, and activity and participation levels in children with DCD.

The hypotheses on which the study proposal is based are as follows:

1. H0: VR application has no effect on motor skills in children with DCD. H1: VR application has an effect on motor skills in children with DCD.
2. H0: VR application has no effect on cognitive skills in children with DCD. H1: VR application has an effect on cognitive skills in children with DCD.
3. H0: VR application has no effect on sensory-perception skills in children with DCD.

   H1: VR application has an effect on sensory-perception skills in children with DCD.
4. H0: VR application has no effect on the functional independence levels in daily living activities in children with DCD.

   H1: VR application has an effect on the functional independence levels in daily living activities in children with DCD.
5. H0: VR application has no effect on participation levels in children with DCD. H1: VR application has an effect on participation levels in children with DCD.

DETAILED DESCRIPTION:
Within the scope of our aims;

* To determine the gross motor skill levels of children with DCD and to obtain the effect of VR application on gross motor skill levels.
* To determine the executive function skill levels of children with DCD and to obtain the effect of VR application on executive function skill levels.
* To determine the sensory-perception skill levels of children with DCD and to obtain the effect of VR application on sensory-perception skill levels.
* To determine the functional independence of children with DCD in daily life and to obtain the effect of VR application on their functional independence levels.
* It is aimed to determine the participation levels of children with DCD and to obtain the effect of VR application on their participation levels.

ELIGIBILITY:
Inclusion Criteria:

* Being between 5-8 years old,
* It is to get 15-46 points from the Developmental Coordination Disorder Questionnaire for ages 5-7 and 15-55 points for ages 8.

Exclusion Criteria:

* Those who are receiving any other therapy program,
* have vision (other than glasses) or hearing problems,
* Children with any neurological disorder will not be included in the study.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Test of Gross Motor Development-2 | It will be applied 8 weeks after the first evaluations are made.
  Assessment of gross and fine motor skills
Sensory İntegration and praxis test | It will be applied 8 weeks after the first evaluations are made.
  It is a standardized test developed by Ayres that evaluates in detail sensory perception and sensory perception-related skills in children between the ages of 4 and 8 years and 11 months. SIPT consists of a total of 17 subtests.
Motor-Free Visual Perception Test-3 | It will be applied 8 weeks after the first evaluations are made.
  Assessment of visual perception

SECONDARY OUTCOMES:
Participation and Environment Measure for Children and Youth (PEM-CY) | It will be applied 8 weeks after the first evaluations are made.
  The PEM-CY is a measure that evaluates participation in the home, at school, and in the community, alongside environmental factors within each of these settings.
CHILDHOOD EXECUTIVE FUNCTIONING INVENTORY (CHEXI) FOR PARENTS AND TEACHERS | It will be applied 8 weeks after the first evaluations are made.
  Working memory and inhibitory control levels will be evaluated with CHEXI.
Functional Independence Measure for Children (WeeFIM) | It will be applied 8 weeks after the first evaluations are made.
  functional independence was assessed with the Functional Independence Measure for Children (WeeFIM).

CONTACTS AND LOCATIONS:
Overall Officials: zeynep kolit, MSc, Principal Investigator — Hacettepe University; Sedef şahin, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)